CLINICAL TRIAL: NCT07277270
Title: A Phase 1b/2 Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Clinical Activity of GSK5764227 in Combination With Standard of Care (SoC) or Other Agents in Participants With Advanced Solid Tumors
Brief Title: A Study of GSK5764227 in Combination With Standard of Care (SoC) or Other Agents in Participants With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 300148; 2025-522274-37-00 (EU CTIS Number)
Record Dates: First submitted 2025-12-02; First posted 2025-12-11 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Neoplasms
Keywords: Solid Tumors; Metastatic colorectal cancer; Metastatic castration-resistant prostate cancer; GSK5764227; Bevacizumab; Fluorouracil; Folinic acid; Enzalutamide; EMBOLD; EMBOLD PanTumor-102
MeSH Terms: conditions — Neoplasms; Colorectal Neoplasms | interventions — Bevacizumab; Fluorouracil; Leucovorin; enzalutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Metastatic colorectal cancer (mCRC) cohort A1 (Experimental)
  Interventions: Drug: GSK5764227; Drug: Bevacizumab
- Metastatic colorectal cancer (mCRC) cohort A2 (Experimental)
  Interventions: Drug: GSK5764227; Drug: Bevacizumab; Drug: Fluorouracil; Drug: leucovorin
- Metastatic castration-resistant prostate cancer (mCRPC) cohort B (Experimental)
  Interventions: Drug: GSK5764227; Drug: Enzalutamide

INTERVENTIONS:
Drug: GSK5764227 — Participants will receive GSK5764227.
Drug: Bevacizumab — Participants will receive bevacizumab.
  Arms: Metastatic colorectal cancer (mCRC) cohort A1; Metastatic colorectal cancer (mCRC) cohort A2
Drug: Fluorouracil — Participants will receive fluorouracil.
  Arms: Metastatic colorectal cancer (mCRC) cohort A2
Drug: leucovorin — Participants will receive leucovorin.
  Arms: Metastatic colorectal cancer (mCRC) cohort A2
Drug: Enzalutamide — Participants will receive enzalutamide.
  Arms: Metastatic castration-resistant prostate cancer (mCRPC) cohort B

SUMMARY:
The goal of this clinical trial is to test a new medicine called GSK5764227, which delivers a toxin directly to cancer cells to destroy them while sparing healthy cells. The study will combine GSK5764227 with standard treatments to evaluate its safety, examine how the body processes it, check if it triggers any immune responses, and assess whether it can shrink or control cancer.

ELIGIBILITY:
Inclusion Criteria:

* Has an ECOG performance status of 0 or 1, with no deterioration in the 2 weeks before first dose.
* Has adequate organ function.
* Has histologically confirmed unresectable adenocarcinoma or unresectable metastatic adenocarcinoma of the colon or rectum. (Cohort A)
* Histologically or cytologically confirmed adenocarcinoma of the prostate (Cohort B)

Exclusion Criteria:

* Has a malignancy (except disease under study) that has progressed or required active treatment within the past 24 months except for basal cell or squamous cell carcinomas of the skin or in-situ carcinomas [e.g., breast, cervix, bladder] that have been resected with no evidence of disease.
* Has had any major surgery within 28 days prior to first dose.
* Has clinically significant bleeding symptoms or significant bleeding tendency within 1 month prior to the first dose.
* Has serious infection within 4 weeks prior to the first dose,
* Has untreated brain or central nervous system (CNS) metastases or brain/CNS metastases that have progressed
* Any evidence of current interstitial lung disease (ILD) or pneumonitis OR a prior history of ILD requiring high-dose glucocorticoids or non-infectious pneumonitis requiring high-dose glucocorticoids.
* Has a history of autoimmune disease that has required systemic treatments in the 2 years prior to screening.
* Has received immunosuppressive agents within 30 days prior to first dose of study intervention (or requires long-term [30 days or longer]). Low-dose corticosteroids (prednisone ≤10 milligrams (mg)/day or equivalent) may be administered.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2025-12-03 (Actual); Primary Completion 2026-07-13 (Estimated); Study Completion 2028-09-29 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events (AEs), Serious AEs (SAEs), AE of special interest (AESIs) and AEs leading to dose modifications | Up to approximately 31 weeks
Number of participants with AEs, SAEs, AESIs, and AEs leading to dose modifications by severity | Up to approximately 31 weeks
Number of participants with dose limiting toxicities (DLTs) | Up to approximately 31 weeks
Number of participants with clinically significant changes in Vital Signs, Body Weight, Laboratory Tests [Hematology, Clinical Chemistry, Urinalysis], Cardiac Function [ECG], and Eastern Cooperative Oncology Group (ECOG) performance status | Up to approximately 31 weeks

SECONDARY OUTCOMES:
Plasma concentration of GSK5764227 [conjugated antibody and payload (GSK5757810) | Up to approximately 112 weeks
Number of participants with anti-drug antibody (ADA) against GSK5764227 | Up to approximately 112 weeks
Number of participants with neutralising antibody (NAb) against GSK5764227 | Up to approximately 112 weeks
Titer of ADA against GSK5764227 | Up to approximately 112 weeks
Objective Response Rate (ORR) | Up to approximately 112 weeks
  ORR is defined as the proportion of participants who have achieved best observed response (BOR) of confirmed complete response (CR) or partial response (PR) as assessed by investigator, according to Response Evaluation Criteria in Solid Tumors (RECIST 1.1) for Cohort A or per Prostate Cancer Clinical Trials Working Group 3 (PCWG3) for Cohort B.
Disease control Rate (DCR18) | Up to approximately 112 weeks
  DCR18 is defined as the proportion of participants who have achieved CR or PR, or stable disease (SD) of ≥17 weeks as assessed by investigator according to PCWG3 for Cohort B.
Duration of Response (DoR) | Up to approximately 112 weeks
  DOR is defined as the time from the date of the first documented objective response (CR/PR) as assessed by investigator according to RECIST 1.1 for cohort A or PCWG3 for cohort B, until the date of the first documented disease progression (PD) or death due to any cause, whichever is earlier.
Progression free survival (PFS) | Up to approximately 112 weeks
  PFS is defined as the time from the date of first dose until the earliest date of documented disease progression as assessed by investigator according to RECIST 1.1 for cohort A.
Radiographic progression-free survival (rPFS) | Up to approximately 112 weeks
  rPFS is defined as the time from the date of first dose until the earliest date of documented PD per PCWG3-modified RECIST 1.1 (soft tissue lesion assessment) and/or PCWG3 bone lesion assessment for cohort B or death due to any cause.
Prostate-specific antigen 50 (PSA50) | Up to approximately 112 weeks
  PSA50 is defined as percentage of participants with a decrease of >=50% in the PSA concentration from the baseline PSA value, confirmed at least 3 weeks later (cohort B)

CONTACTS AND LOCATIONS:
Locations (5):
- GSK Investigational Site, Lake Success, New York, United States
- GSK Investigational Site, Tugun, Queensland, Australia
- Spain (3):
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Málaga

IPD SHARING:
Plan to Share IPD: Yes
Study Sponsor will assess requests from qualified researchers for anonymized individual patient-level data and related study documents. Data sharing is subject to certain criteria, conditions, and exceptions. For further information, refer to https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or asset(s) with development terminated across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months, but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf